CLINICAL TRIAL: NCT06741254
Title: The Effect of Stress Ball on Anxiety, Comfort and Non Stress Test Parameters of Pregnant Women During Non Stress Testing: A Randomized Controlled Trial
Brief Title: The Effect of Stress Ball on Anxiety, Comfort and Non Stress Test Parameters of Pregnant Women During Non Stress Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zehra Çerçer, Assistant Professor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/444
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Comfort
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Stress Ball) (Experimental): Pregnant women included in the experimental group will be asked for written informed consent before the NST application, and the Pregnant Descriptive Information Form, State Anxiety Scale and Visual Comfort Scale will be completed. Then, the NST device will be connected to the pregnant woman and the Stress ball application will be started. During the NST procedure (average 20-30 minutes), the pregnant woman will lie on her left side. A stress ball will be placed in the right hand of the pregnant woman. The pregnant woman will be instructed to squeeze the stress ball for 2-3 seconds and then relax the hand and arm. This process will be repeated throughout the NST. During the NST application, the pregnant researcher will remain under the supervision of the midwife/nurse. The State Anxiety Scale and Visual Comfort Scale will be repeated immediately after the NST procedure. The NST result form will be filled out according to the NST printout.
  Interventions: Other: Stress Ball
- Control (No Intervention): Written informed consent will be obtained from the pregnant women in the control group before the NST application, and the Pregnant Descriptive Information Form, State Anxiety Scale and Visual Comfort Scale will be completed. Then the NST device will be connected to the pregnant woman. Pregnant women in this group will not be given a stress ball. During the NST procedure (average 20-30 minutes), the pregnant woman will lie on her left side. During the NST procedure, the pregnant woman will remain under the supervision of the researcher midwife/nurse. The State Anxiety Scale and Visual Comfort Scale will be repeated immediately after the NST procedure. The NST result form will be filled according to the NST trace.

INTERVENTIONS:
Other: Stress Ball — During the NST procedure (average 20-30 minutes), the pregnant woman will lie on her left side. A stress ball will be placed in the right hand of the pregnant woman. The pregnant woman will be instructed to squeeze the stress ball for 2-3 seconds and then relax the hand and arm. This process will be repeated throughout the NST.
  Arms: Experimental (Stress Ball)

SUMMARY:
Non-stress testing (NST) is used to assess fetal wellbeing and to detect and intervene early in fetuses at risk. NST is an easy to administer, noninvasive, prenatal assessment method used from 32 weeks of gestation to term. High levels of anxiety during the common NST procedure can negatively affect the test result and increase the rate of nonreactive NST, potentially leading to misinterpretation. Therefore, midwifery/nursing interventions to make the pregnant woman comfortable during the procedure and to reduce anxiety and stress are important.

DETAILED DESCRIPTION:
Non-stress testing (NST) is used to assess fetal wellbeing and to detect and intervene early in fetuses at risk. NST is an easy to administer, noninvasive, prenatal assessment method used from 32 weeks of gestation to term. High levels of anxiety during the common NST procedure can negatively affect the test result and increase the rate of non-reactive NST, potentially leading to misinterpretation. Therefore, midwifery/nursing interventions to make the pregnant woman comfortable during the procedure and to reduce anxiety and stress are important. Stress ball is one of the nonpharmacological methods in the management of pain, stress and anxiety based on the logic of drawing the attention of the person to a different side and is an application for the sense of touch. In the obstetric field, there have been studies evaluating the effects of stress ball application on labor and vascular pain of pregnant women, but there is no study evaluating anxiety, comfort and NST parameters during NST.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-35,
* Turkish as the mother tongue,
* Being literate, having a singleton pregnancy,
* She has had NST at least once before,
* 32 weeks or more gestation,
* Being multiparous,
* Having eaten at least two hours before the NST procedure,
* Volunteering to participate in the research.

Exclusion Criteria:

* Having a high-risk pregnancy,
* Having a psychiatric disorder,
* Being pregnant with an urgent NST result,
* Smoking or drinking alcohol at least two hours before the NST procedure,
* Having any problem that prevents communication (such as hearing, speaking, ability to understand), having a visual, hearing, speech, physical or mental disability.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | 1 minute before NST application and 1 minute after NST aplication
  The scale was created by Spielberger. Its Turkish validity and reliability was performed by Öner and Le Compte. It is a 4-point Likert-type scale consisting of 20 questions measuring the anxiety levels of individuals. The scale includes items that are expressed positively and negatively. In the scoring phase of the scale, the total weighted score obtained for the direct statements is subtracted from the total weighted score of the reversed statements. A predetermined and unchanging value is added to this number. This unchanging value is 50 for the State Anxiety Scale. The last value obtained gives the anxiety score of the person. The scores that can be obtained from the scale vary between 20 and 80, and high scores indicate a high level of anxiety. The Cronbach alpha value of the original scale is between 0.94-0.96 and has a high internal consistency.

SECONDARY OUTCOMES:
Visual Analog Scale for Comfort | 1 minute before NST application and 1 minute after NST aplication
  The Visual Analog Scale (VAS) is a reliable, valid and sensitive self-report measure for the examination of subjective patient experiences including pain, nausea, fatigue and dyspnea.The VAS scale consists of 0-10 points. Pregnant women will be asked to mark a number according to the comfort they feel. A score of '0' indicates feeling uncomfortable, while a score of '10' indicates the highest level of comfort.

OTHER OUTCOMES:
NST Result Form | 1 minute after NST aplication
  This form was created by utilizing the literature. In the form, 6 criteria including basal fetal heart rate, number of fetal movements, variability (present/absent), number of accelerations, number of contractions (40 mm/Hg and above) and reactivity in NST interpretation (reactive/nonreactive) will be evaluated. Reactive NST; The test result will be considered as reactive NST if the electronic fetal heart rate tracing recorded in a 20 minute time period has at least two accelerations lasting at least 15 seconds and 15 beats/minute more than the initial beat. Nonreactive NST; The test result will be considered nonreactive NST if the electronic fetal heart rate trace recorded during the 20 minute time period does not have at least two accelerations lasting at least 15 seconds and at least 15 beats/minute greater than the baseline beat.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra ÇERÇER, PhD, Principal Investigator — Gaziantep Islam Science Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toker E, Gokduman Keles M. The effect of virtual reality on fetal movement, fetal heart rate, maternal satisfaction, fatigue, and anxiety levels and vital signs of pregnant women during non-stress test: A randomized controlled trial. Health Care Women Int. 2024;45(7):765-781. doi: 10.1080/07399332.2023.2223159. Epub 2023 Jun 22. PMID 37347556
- [Background] Yilmaz Sezer N, Aker MN, Yucel A, Calisici D. The effect of virtual reality and music on anxiety, non-stress test parameters, and satisfaction of high-risk pregnant women undergoing non-stress tests: Randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2024 May;296:52-58. doi: 10.1016/j.ejogrb.2024.02.038. Epub 2024 Feb 21. PMID 38394716
- [Background] Hobek Akarsu R, Kus B, Dogukan Akarsu G. Effects of Valsalva Maneuver, EMLA Cream, and Stress Ball for Pregnant Women's Venipuncture Pain. Altern Ther Health Med. 2021 Sep;27(5):108-114. PMID 33626021